CLINICAL TRIAL: NCT00623766
Title: A Multi-Center Phase II Study to Evaluate Tumor Response to Ipilimumab (BMS-734016) Monotherapy in Subjects With Melanoma Brain Metastases
Brief Title: Evaluation of Tumor Response to Ipilimumab in the Treatment of Melanoma With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-042
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ipilimumab, 10 mg/kg, IV in corticosteroid-free patients (Experimental): Participants who had not received corticosteroid therapy for at least 10 days before starting study drug received ipilimumab,10 mg/kg, as a 90-minute intravenous (IV) infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV, every 12 weeks, beginning at Week 24.
  Interventions: Drug: Ipilimumab
- Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients (Experimental): Participants who were dependent on corticosteroid therapy received ipilimumab, 10 mg/kg, as a 90-minute intravenous (IV) infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV, every 12 weeks, beginning at Week 24.
  Interventions: Drug: Ipilimumab; Drug: Corticosteroid: Betamethasone; Drug: Corticosteroid: Dexamethasone; Drug: Corticosteroid: Fludrocortisone; Drug: Corticosteroid: Hydrocortisone; Drug: Corticosteroid: Meprednisone; Drug: Corticosteroid: Methylprednisolone; Drug: Corticosteroid: Prednisolone; Drug: Corticosteroid: Prednisone; Drug: Corticosteroid: Triamcinolone

INTERVENTIONS:
Drug: Ipilimumab — 10 mg/kg, administered as an intravenous infusion every 3 weeks during induction and every 12 weeks during maintenance
  Other Names: BMS-734016; MDX-010
Drug: Corticosteroid: Betamethasone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with betamethasone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Dexamethasone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with dexamethasone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Fludrocortisone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with fludrocortisone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Hydrocortisone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with hydrocortisone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Meprednisone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with meprednisone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Methylprednisolone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with methylprednisolone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Prednisolone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with prednisolone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Prednisone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with prednisone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients
Drug: Corticosteroid: Triamcinolone — Participants in the corticosteroid-dependent arm for whom adequate control of metastatic brain lesion-related neurologic signs and symptoms required concurrent corticosteroid therapy with triamcinolone
  Arms: Ipilimumab, 10 mg/kg, IV in corticosteroid-dependent patients

SUMMARY:
To assess the response of melanoma with brain metastases to ipilimumab treatment while maintaining acceptable tolerability.

ELIGIBILITY:
Key inclusion criteria

* Histologically confirmed malignant melanoma
* At least 1 measurable index brain metastasis >0.5 cm and no larger than 3 cm in diameter that had not been previously irradiated, and/or 2 measurable lesions >0.3 cm visible on contrast magnetic resonance
* Index brain lesion must have resolved consequences of prior therapy that could have confounded attribution of tumor response including edema and hemorrhage
* Participants in ipilimumab monotherapy arm (including the first 21 who were enrolled in Stage 1) were to be free of neurologic symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroid therapy in the 10 days prior to beginning ipilimumab therapy
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Required values for initial laboratory tests:

  * White blood cell count ≥2000/μL
  * Absolute neutrophil count ≥1000/μL
  * Platelets ≥100*10^3/μL
  * Hemoglobin level ≥9 g/dL (may have been transfused)
  * Aspartate aminotransferase/alanine aminotransferase (AST/ALT) level ≤2.5*ULN for participants without liver metastasis
  * AST/ALT level ≤5*ULN for those with liver metastasis
  * Bilirubin level ≤2*ULN (except participants with Gilbert's Syndrome, who must have had a total bilirubin level less than 3.0 mg/dL)
* Age 16 years and older
* Males and females
* Women of childbearing potential (WOBP) must be using an adequate method of contraception to avoid pregnancy throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal.

Key exclusion criteria

* History of carcinomatous meningitis, with prior stereotactic or highly conformal radiotherapy and/or whole brain irradiation within 14 days before the first dose of ipilimumab, and documented history of autoimmune disease
* Prior stereotactic or highly conformal radiotherapy and/or whole brain irradiation within 14 days prior to start of ipilimumab dosing for this study. Note the stereotactic radiotherapy field must not have included the brain index lesion or the lesion must have been detected and confirmed to be active and progressing after receiving whole brain irradiation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City Of Hope, Duarte, California
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution, The Bronx, New York
  - Providence Portland Med Ctr, Portland, Oregon
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Derived] Johnson DB, Friedman DL, Berry E, Decker I, Ye F, Zhao S, Morgans AK, Puzanov I, Sosman JA, Lovly CM. Survivorship in Immune Therapy: Assessing Chronic Immune Toxicities, Health Outcomes, and Functional Status among Long-term Ipilimumab Survivors at a Single Referral Center. Cancer Immunol Res. 2015 May;3(5):464-9. doi: 10.1158/2326-6066.CIR-14-0217. Epub 2015 Feb 3. PMID 25649350
- [Derived] Iwama S, De Remigis A, Callahan MK, Slovin SF, Wolchok JD, Caturegli P. Pituitary expression of CTLA-4 mediates hypophysitis secondary to administration of CTLA-4 blocking antibody. Sci Transl Med. 2014 Apr 2;6(230):230ra45. doi: 10.1126/scitranslmed.3008002. PMID 24695685
- [Derived] Margolin K, Ernstoff MS, Hamid O, Lawrence D, McDermott D, Puzanov I, Wolchok JD, Clark JI, Sznol M, Logan TF, Richards J, Michener T, Balogh A, Heller KN, Hodi FS. Ipilimumab in patients with melanoma and brain metastases: an open-label, phase 2 trial. Lancet Oncol. 2012 May;13(5):459-65. doi: 10.1016/S1470-2045(12)70090-6. Epub 2012 Mar 27. PMID 22456429
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 99 participants were enrolled, and 27 did not receive treatment because they did not meet screening criteria.
Groups:
- Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients: Participants who had not received corticosteroid therapy for at least 10 days before starting study drug received ipilimumab,10 mg/kg, as a 90-minute intravenous (IV) infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV every 12 weeks, beginning at Week 24.
- Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients: Participants who required concurrent systemic corticosteroid therapy for adequate control of neurologic signs and symptoms related to metastatic brain lesion received ipilimumab,10 mg/kg, as a 90-minute IV infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV every 12 weeks, beginning at Week 24.
Period: Induction Phase (Day 1 to Week 24)
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Started | 51 (Participants who received treatment) | 21 (Participants who received treatment)
Completed | 15 (4 patients completed Induction but did not enter Maintenance; they were only followed up with scans.) | 5 (3 patients completed Induction but did not enter Maintenance; they were only followed up with scans.)
Not Completed | 36 | 16
Not completed — Off treatment | 36 | 16
Period: Maintenance Phase (Week 24 to Year 2)
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Started | 11 | 2
Completed | 1 (Inadvertently not noted as discontinued (disease progression); data collection error at site closure) | 0
Not Completed | 10 | 2
Not completed — Disease progression | 4 | 0
Not completed — Administrative reason by sponsor | 4 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Patient required surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients: Participants who were dependent on corticosteroid therapy received ipilimumab,10 mg/kg, as a 90-minute IV infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV every 12 weeks, beginning at Week 24.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients | Total
Number analyzed (Participants) | 51 | 21 | 72
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 39 | 17 | 56
  65 years and older | 12 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 33 | 11 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 51 | 21 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) score [Number; unit: Units on a scale] — ECOG performance status assesses a participant's physical ability on a 6-point scale: 0=fully active, able to carry on all predisease activities without restriction; 1=restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Score of 0=best status and 5=worst status.
  Units on a scale
    0 | 25 | 14 | 39
    1 | 26 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate by Modified World Health Organization (mWHO) Tumor Assessment Criteria
Description: Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) (global, in brain, or outside of brain) based on mWHO criteria divided by the number of patients who received treatment. By mWHO criteria: CR=complete disappearance of all index lesions. PR=decrease, relative to baseline, of 50% or greater in the sum of the 2 largest perpendicular diameters of all index lesions. SD=does not meet criteria for CR or PR, in the absence of progressive disease (PD). Patients with PR or CR not confirmed after at least 4 weeks are scored as SD unless they have new primary lesions. PD=at least 25% increase in the sum of the diameters of all index lesions (taking as reference the smallest sum recorded at or following baseline) and/or the appearance of any new lesions. CNS=central nervous system.
Time Frame: From Day 1, first dose to end of Week 12
Population: All participants who received at least 1 dose of ipilimumab
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Percentage of participants
  Global disease control rate | 17.6 [8.4 to 30.9] | 4.8 [0.1 to 23.8]
  Disease control rate in brain | 23.5 [12.8 to 37.5] | 9.5 [1.2 to 30.4]

2. Secondary Outcome: Disease Control Rate by Immune-related Response Criteria (irRC)
Description: Disease control rate is defined as the number of patients with a best overall response of immune-related (ir) complete response (irCR), partial response (irPR), or stable disease (irSD) divided by the total number of patients who received treatment. By irRC definition: irCR=complete disappearance of all index lesions. irPR=decrease, relative to baseline, of 50% or greater in the sum of the products of the 2 largest perpendicular diameters of all index lesions. irSD=does not meet criteria for irCR or irPR, in the absence of ir progressive disease (irPD). irPD=at least 25% increase in the sum of the products of all index lesions (taking as reference the smallest sum recorded at or following baseline). CNS=central nervous system; non-CNS compartment=extracranial, or outside of the brain.
Time Frame: From Day 1, first dose to end of Week 12
Population: All participants who received at least 1 dose of ipilimumab
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Ipilimumab 10 mg/kg IV, in Corticosteroid-free Patients: Participants who had not received corticosteroid therapy for at least 10 days before starting study drug received ipilimumab,10 mg/kg, as a 90-minute intravenous (IV) infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV every 12 weeks, beginning at Week 24.
Arm/Group | Ipilimumab 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Percentage of participants
  Global disease control rate | 25.5 [14.3 to 39.6] | 9.5 [1.2 to 30.4]
  Disease control rate in brain lesions | 25.5 [14.3 to 39.6] | 9.5 [1.2 to 30.4]
  Disease control rate in non-CNS compartment | 33.3 [20.8 to 47.9] | 9.5 [1.2 to 30.4]

3. Secondary Outcome: Best Overall Response Rate (BORR) by Modified World Health Organization (mWHO) Criteria and by Immune-relate Response Criteria (irRC)
Description: BORR is defined as the number of patients whose global best overall response (BOR) was complete (CR) or partial response (PR), divided by the total number of participants who received treatment. CR=complete disappearance of all index lesions. PR=decrease, relative to baseline, of 50% or greater in the sum of the products of the 2 largest perpendicular diameters of all index lesions. The global BOR is the best overall response (OR) designation over the study as a whole for an individual in the study based on overall tumor burden. Both central nervous system (CNS) (brain lesions) and non-CNS compartments (lesions outside the brain) are considered for the global BOR. For the analysis of global BOR of CR or PR (by both modified WHO criteria and immune-related response criteria [irRC]), the OR assessment must be confirmed by a second (confirmatory) evaluation meeting the criteria for response and must be performed no less than 4 weeks after the criteria for response are first met.
Time Frame: From Day 1, first dose until the last tumor assessment, Week 12
Population: All participants who received at least 1 dose of ipilimumab
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Percentage of participants
  Global BORR (mWHO criteria) | 9.8 [3.3 to 21.4] | 4.8 [0.1 to 23.8]
  BORR in brain (mWHO criteria) | 15.7 [7.0 to 28.6] | 4.8 [0.1 to 23.8]
  BORR in non-CNS compartment (mWHO criteria) | 13.7 [5.7 to 26.3] | 4.8 [0.1 to 23.8]
  Global BORR (irRC) | 9.8 [3.3 to 21.4] | 4.8 [0.1 to 23.8]
  BORR in brain (irRC) | 15.7 [7.0 to 28.6] | 4.8 [0.1 to 23.8]
  BORR in non-CNS compartment (irRC criteria ) | 13.7 [5.7 to 26.3] | 4.8 [0.1 to 23.8]

4. Secondary Outcome: Duration of Response (DOR) by Modified World Health Organization (mWHO) Criteria and by Immune-related Response Criteria (irRC)
Description: DOR is defined in patients whose global best overall response is complete (CR) or partial response (PR) as the time between the date of response of confirmed CR or PR, whichever occurs first, and the date of progressive disease or death, whichever occurs first. For patients who remain alive and have not progressed following response, duration of response will be censored on the date of last evaluable tumor assessment.
Time Frame: From Day 1, first dose to last tumor assessment up to 18.2 months
Population: All participants who received at least 1 dose of ipilimumab
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Months
  DOR by mWHO criteria | 10.4 [2.9 to 18.2] | NA [NA to NA] — The only corticosteroid-dependent patient with response has not progressed or died
  DOR by irRC | 10.4 [2.9 to 18.2] | NA [NA to NA] — The only corticosteroid-dependent patient with response has not progressed or died

5. Secondary Outcome: Progression-free Survival (PFS) by Modified World Health Organization (mWHO) Criteria and by Immune-related Response Criteria (irRC)
Description: PFS is defined as the time between the date of the first dose of study therapy and the date of progression or death, whichever occurs first. A patient who dies without reported prior progression will be considered to have progressed on the date of death. For those who remain alive and have not progressed, PFS will be censored on the date of last evaluable tumor assessment. Participants who have not died and have no recorded postbaseline tumor assessment will be censored on the date of first dose of study therapy. Those who die without any recorded postbaseline tumor assessment will be considered to have progressed on the date of death.
Time Frame: From Day 1, first dose to the date of progression or death, whichever occurred first up to 22 months
Population: All participants who received at least 1 dose of ipilimumab
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Months
  Global PFS (mWHO criteria) | 1.4 [1.2 to 2.6] | 1.2 [1.2 to 1.3]
  PFS in brain (mWHO criteria) | 1.5 [1.2 to 2.6] | 1.2 [1.2 to 1.3]
  PFS in non-CNS compartment (mWHO criteria) | 2.6 [1.3 to 4.1] | 1.3 [1.2 to 2.5]
  Global PFS (irRC) | 2.7 [1.6 to 3.7] | 1.3 [1.2 to 2.5]
  PFS in brain (irRC) | 1.9 [1.2 to 2.9] | 1.2 [1.2 to 1.3]
  PFS in non-CNS compartment (irRC) | 3.3 [2.6 to 4.7] | 1.3 [1.2 to 2.5]

6. Secondary Outcome: Number of Participants Surviving at 6, 12, 18, 24, and 36 Months (Overall Survival [OS] Rate)
Description: OS is defined as the time from the first dose of study drug until the date of death. Overall survival rate is the percentage of participants known to be alive at a timepoint. For those patients who did not die, OS was censored at the recorded last date of patient contact, and those with a missing recorded last date of contact will be censored at the last date the patient was known to be alive. The survival rate at a specified time-point is the probability that a patient is alive at that time following randomization. The rate is calculated for each treatment group using the Kaplan-Meier product-limit method. A corresponding 2-sided 95% bootstrap confidence interval will be calculated.
Time Frame: From first dose to Months 6, 12, 18, 24, and 36 months
Population: All participants who received at least 1 dose of ipilimumab
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Probability of being alive
  At 6 months | 0.55 [0.41 to 0.68] | 0.38 [0.17 to 0.59]
  At 12 months | 0.31 [0.18 to 0.44] | 0.19 [0.02 to 0.36]
  At 18 months | 0.26 [0.14 to 0.39] | 0.19 [0.02 to 0.36]
  At 24 months | 0.26 [0.14 to 0.39] | 0.10 [0.00 to 0.22]
  At 36 months | 0.26 [0.14 to 0.39] | 0.10 [0.00 to 0.22]

7. Secondary Outcome: Number of Participants Who Died or Had a Treatment-related Adverse Event (AE), Immune-related AE, Immune-related Serious Adverse Event (SAE), Nervous System Disorder, Treatment-related Nervous System Disorder, SAE, and AE Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: Continuously from Day 1, first dose, to 70 days following last dose of ipilimumab
Population: All participants who received at least 1 dose of ipilimumab
Measure: Number; unit: Participants
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Participants
  Deaths | 37 | 20
  Treatment-related AEs (all) | 45 | 17
  Treatment-related AEs (Grade 3/4) | 17 | 4
  Treatment-related AEs (Fatal) | 0 | 0
  Immune-related AEs (All) | 35 | 13
  Immune-related AEs (Grade 3/4) | 11 | 3
  Immune-related AEs (Fatal) | 0 | 0
  Immune-related SAEs (All) | 11 | 6
  Immune-related SAES (Grade 3/4) | 7 | 3
  Immune-related SAES (Fatal) | 0 | 0
  Nervous system disorder (NSD) (All) | 40 | 14
  NSD (Grade 3/4) | 17 | 7
  NSD (Fatal) | 0 | 1
  Treatment-related NSD (All) | 8 | 3
  Treatment-related NSD (Gr 3/4) | 1 | 0
  Treatment-related NSD (Fatal) | 0 | 0
  SAE (All) | 36 | 17
  SAE (Grade 3/4) | 18 | 7
  SAE (Fatal) | 17 | 10
  AEs leading to discontinuation (All) | 15 | 9
  AEs leading to discontinuation (Grade 3/4) | 9 | 4
  AEs leading to discontinuation (Fatal) | 5 | 4

8. Secondary Outcome: Onset of Response by Modified World Health Organization (mWHO) Criteria and Immune-related Response Criteria (irRC)
Description: Onset of response is defined as the time between the first dose of study therapy and the date when measurement criteria are first met for global best overall response of partial (PR) or complete (CR), whichever occurs first. CR=complete disappearance of all index lesions. PR=decrease, relative to baseline, of 50% or greater in the sum of the 2 largest perpendicular diameters of all index lesions.
Time Frame: From Day 1, first dose to a maximum of 4.2 months
Population: All participants who received at least 1 dose of ipilimumab. n=number of participants with a best overall response of CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Months
  Onset of response (mWHO criteria) (n=5, 1) | 1.2 [1.1 to 4.2] | 1.2 [1.2 to 1.2]
  Onset of response (irRC) (n=5, 1) | 1.2 [1.1 to 4.2] | 1.2 [1.2 to 1.2]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of first dose of study drug until the date of death. For those patients who did not die, OS was censored at the recorded last date of patient contact, and those missing a recorded last date of contact will be censored at the last date the patient was known to be alive.
Time Frame: From first dose to 24 months
Population: All participants who received at least 1 dose of ipilimumab
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ipilimumab, 10 mg/kg, IV in Corticosteroid-dependent Patients: Participants who required concurrent systemic corticosteroid therapy for adequate control of neurologic signs and symptoms related to metastatic brain lesion received ipilimumab,10 mg/kg, as a 90-minute IV infusion every 3 weeks (Weeks 1, 4, 7, and 10) during the Induction Phase. Those eligible (patients who did not discontinue due to toxicity, did not show progression at 24 weeks, and who remained clinically stable) for the Maintenance Phase continued to receive ipilimumab, 10 mg/kg IV every 12 weeks, beginning at Week 24.
Arm/Group | Ipilimumab, 10 mg/kg, IV in Corticosteroid-free Patients | Ipilimumab, 10 mg/kg, IV in Corticosteroid-dependent Patients
Number analyzed (Participants) | 51 | 21
Months | 6.97 [4.14 to 10.81] | 3.75 [1.64 to 7.33]

ADVERSE EVENTS:
Arm/Group | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients
Serious Adverse Events (participants affected / at risk) | 17/21 | 36/51
Other Adverse Events (participants affected / at risk) | 20/21 | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients (N=21) | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients (N=51)
Ataxia (Nervous system disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 3
Fatigue (General disorders) | 1 | 2
Pyrexia (General disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Pneumonia viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Disease progression (General disorders) | 10 | 16
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 6
Headache (Nervous system disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 2
Aphasia (Nervous system disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Colon gangrene (Infections and infestations) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 2 | 5
Depressed level of consciousness (Nervous system disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 5
Alanine aminotransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 5
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Convulsion (Nervous system disorders) | 3 | 3
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 5
Pain (General disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, 10 mg/kg IV, in Corticosteroid-dependent Patients (N=21) | Ipilimumab, 10 mg/kg IV, in Corticosteroid-free Patients (N=51)
Fatigue (General disorders) | 11 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pyrexia (General disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 7 | 20
Dizziness (Nervous system disorders) | 2 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Haemoglobin decreased (Investigations) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Influenza like illness (General disorders) | 0 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 0
Visual impairment (Eye disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 14
Dysgeusia (Nervous system disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Herpes zoster (Infections and infestations) | 0 | 3
Insomnia (Psychiatric disorders) | 4 | 8
Paraesthesia (Nervous system disorders) | 3 | 1
Thirst (General disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 3
Brain oedema (Nervous system disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 5 | 9
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 24
Headache (Nervous system disorders) | 6 | 20
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3
Memory impairment (Nervous system disorders) | 0 | 5
Oedema peripheral (General disorders) | 6 | 4
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Weight decreased (Investigations) | 1 | 7
Adrenal insufficiency (Endocrine disorders) | 2 | 1
Aphasia (Nervous system disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 4
Blood alkaline phosphatase increased (Investigations) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Gait disturbance (General disorders) | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3
Polyuria (Renal and urinary disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Confusional state (Psychiatric disorders) | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4
Hypertension (Vascular disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 1 | 10
Alanine aminotransferase increased (Investigations) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Bronchitis (Infections and infestations) | 0 | 3
Chills (General disorders) | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Sinusitis (Infections and infestations) | 0 | 6
Vision blurred (Eye disorders) | 2 | 7
Convulsion (Nervous system disorders) | 1 | 5
Flatulence (Gastrointestinal disorders) | 2 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 4 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.